CLINICAL TRIAL: NCT01470963
Title: Practical Health Co-operation - a Randomised Controlled Intervention Study. The Impact of a Referral Template on Quality of Care and Health Care Co-operation Between Primary and Secondary Care
Brief Title: Practical Health Co-operation - The Impact of a Referral Template on Quality of Health Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: University of Tromso (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HST1026-11
Record Dates: First submitted 2011-09-05; First posted 2011-11-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Referral; Quality of Health Care
Keywords: Referral; Quality of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Referral template (Experimental): Implementation of the referral templates at the GP office
  Interventions: Other: Implementation of referral template
- Control (No Intervention): Normal referral pattern

INTERVENTIONS:
Other: Implementation of referral template — Implementation of referral template at the GP office
  Arms: Referral template

SUMMARY:
The purpose of this study is to examine whether the implementation of a referral template will increase quality of health care delivered and the quality of health care co-operation. The investigators intent to implement a referral template, at the level of the general practitioner (GP), for the referral of patients within 4 separate diagnostic groups:

* dyspepsia/upper GI symptoms
* colonic cancer investigation/lower GI symptoms
* chronic obstructive pulmonary disease (COPD)
* chest pain

Local GP clinics will be randomised to use the referral template or to use standard referral practice. Using a predefined set of quality criteria the investigators will score the process of care in each patient, and compare intervention and control groups. In addition other criteria will be collected and compared between the two groups, e.g.

* time to diagnosis/treatment
* quality of referral
* more appropriate referrals
* patient satisfaction (as measured by a questionnaire)

The investigators hypothesize that the implementation of a referral template will lead to a measurable increase in the quality of health care delivered.

DETAILED DESCRIPTION:
There is a continuous work to improve the quality of health care delivered to an individual patient, both in primary and secondary care. The referral from primary to secondary care represents a key component in the communication between the levels of care, and therefore an important tool in developing the quality of care. There has been many attempts at improving the quality of referrals, but less work has been focussed on the consequence of such improvement on quality of health care. This study is designed as a randomised controlled intervention study where we intent to implement a referral templates, at the level of the general practitioner (GP). These templates will be for the referral of patients within 4 separate diagnostic groups:

* dyspepsia/upper GI symptoms
* colonic cancer investigation/lower GI symptoms
* chronic obstructive pulmonary disease (COPD)
* chest pain

Following the course of the health care process we will assess the quality of the care process by using predefined quality of care criteria, together with patient satisfaction (as measured by questionnaire) and other health process indicators.

Our primary hypothesis is that the implementation of a referral template in the communication between primary and secondary care, will lead to a measurable increase in the quality of health care delivered.

Secondary hypothesis include:

* the use of a referral template in the communication between the GP and secondary care, will lead to better patient satisfaction.
* the use of a referral template in the communication between the GP and secondary care, will lead to a change (up or down) in the amount of patients defined as being in need of prioritisation (as defined pr. national guidelines for prioritisation in health care)
* the use of a referral template in the communication between the GP and secondary care, will lead to a measurable referral quality improvement
* the use of a referral template in the communication between the GP and secondary care, will increase the "appropriateness" of the referrals

ELIGIBILITY:
Inclusion Criteria:

* referral to medical department of University Hospital of North Norway, Harstad

Exclusion Criteria:

* children (< 18 years of age)
* patients with reduced capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2011-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Collated quality indicator score | The care period for each patient (approx. 3 weeks up to 1 year)
  Based on treatment guidelines and international quality assessment tools we have developed quality indicators score sets for each of the 4 diagnostic groups in the study. The scores will be compared between intervention and control GP offices to assess the effect of the referral template.

SECONDARY OUTCOMES:
Improved referral quality | The care period for each patient (approx. 3 weeks up to 1 year)
  The investigators will evaluate each referral against the referral template, and then compare between intervention and control groups.
Waiting time from referral to appointment | The care period for each patient (approx. 3 weeks up to 1 year)
Time from referral to initiation of treatment | The care period for each patient (approx. 3 weeks up to 1 year)
  Compare the time from referral to initiation of treatment/"decision no treatment" necessary between intervention and control groups
Percentage of patients seen within investigation deadline | Assessed at end of study - approx 2 years
  Compare the number of patients in the two groups seen within the limit set in national prioritisation guidelines
Number of patients designated with investigation deadline | Assessed at end of study - approx 2 years
  Compare the number of patients in the intervention vs. control group that were designated with a investigation deadline according to national prioritisation guidelines
Patient satisfaction | The care period for each patient (approx. 3 weeks up to 1 year)
  Patient satisfaction as measured by self report questionnaire
Positive predictive value of referral | The care period for each patient (approx. 3 weeks up to 1 year)
  Compare the percentage of referrals between the intervention and control groups which have lead to
  1. a diagnostic clarification, or
  2. a histological diagnosis, or
  3. a change in medical management
Number of appointments needed for diagnostic clarification | The care period for each patient (approx. 3 weeks up to 1 year)
  Compare the number of appointments needed to clarify diagnosis between intervention and control groups

CONTACTS AND LOCATIONS:
Overall Officials: Ann Ragnhild Broderstad, Dr. med, Principal Investigator — University Hospital of North Norway
Locations (1):
- Medical department - University Hospital of North Norway Harstad, Harstad, Norway

REFERENCES:
- [Derived] Wahlberg H, Valle PC, Malm S, Hovde O, Broderstad AR. The effect of referral templates on out-patient quality of care in a hospital setting: a cluster randomized controlled trial. BMC Health Serv Res. 2017 Mar 7;17(1):177. doi: 10.1186/s12913-017-2127-1. PMID 28270128
- [Derived] Wahlberg H, Braaten T, Broderstad AR. Impact of referral templates on patient experience of the referral and care process: a cluster randomised trial. BMJ Open. 2016 Oct 24;6(10):e011651. doi: 10.1136/bmjopen-2016-011651. PMID 27797992
- [Derived] Wahlberg H, Valle PC, Malm S, Broderstad AR. Impact of referral templates on the quality of referrals from primary to secondary care: a cluster randomised trial. BMC Health Serv Res. 2015 Aug 29;15:353. doi: 10.1186/s12913-015-1017-7. PMID 26318734
- [Derived] Wahlberg H, Valle PC, Malm S, Broderstad AR. Practical health co-operation - the impact of a referral template on quality of care and health care co-operation: study protocol for a cluster randomized controlled trial. Trials. 2013 Jan 7;14:7. doi: 10.1186/1745-6215-14-7. PMID 23295103